CLINICAL TRIAL: NCT01975636
Title: An Open-label, Single Dose Study to Determine the Metabolism and Elimination of [14C]E2609 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2609-A001-005
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-11

CONDITIONS: Metabolism and Elimination
Keywords: Metabolism and Elimination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E2609 (Experimental): Single oral 100 mg +/- 10 mg E2609 with a level of radioactive exposure consistent with the Radioactive Drug Research Committee allowance
  Interventions: Drug: E2609

INTERVENTIONS:
Drug: E2609 — Single oral 100 mg +/- 10 mg E2609 with a level of radioactive exposure consistent with the Radioactive Drug Research Committee allowance

SUMMARY:
This is an open-label, single dose study in healthy male subjects.

DETAILED DESCRIPTION:
A baseline (predose) fecal sample and a baseline (predose) urine sample will be obtained at the clinic prior to dosing on Day 1.

On Day 1, subjects will begin the Treatment Phase. Subjects will be released from the clinic after at least 10 days since dosing and as soon as the following conditions are met:

* greater than 90% of the administered radioactivity has been recovered, and
* less than 1% of the administered radioactive dose is recovered in two consecutive 24-hour samples each of urine and feces

ELIGIBILITY:
Inclusion Criteria

Subjects must meet criteria to be included in this study, including but not limited to the following:

1. Healthy male 18 - 55 years, inclusive, at the time of informed consent
2. Body mass index (BMI) of 18 to 32 kg/m2 at Screening
3. Subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners not be of childbearing potential or must be practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation. Sperm donation is not allowed during the study period and for 30 days after study drug discontinuation.
4. Provide written informed consent
5. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Have participated in a 14C-research study within the 6 months prior to Day -2. The total exposure from this and any previous study must be within the recommended levels considered safe.
2. Exposure to clinically significant radiation within 12 months prior to Day -2.
3. Any laboratory abnormalities considered clinically significant by the investigator, which may require further investigations or treatment
4. Clinically significant illness which required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing
5. Any history of gastrointestinal surgery (e.g., hepatectomy, nephrotomy, digestive organ resection) that may affect PK profiles of study drugs
6. Hypersensitivity to the study drugs or any of their excipients
7. Known to be human immunodeficiency virus (HIV) positive

Restrictions will apply on prior and concomitant medications, food and beverages

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Elimination of E2609: urine/feces concentration | Predose and every 24 hours postdose up to 28 days
  Total radioactivity will be analyzed in urine and feces predose and up to 28 days postdose.
Pharmacokinetics: Plasma concentration of E2609/metabolite | Predose andup to 648 hours postdose
  Total radioactivity will be analyzed in whole blood, plasma, and red blood cells.

SECONDARY OUTCOMES:
Pharmacokinetics: Metabolic profile of E2609: plasma/urine/feces concentration | Predose andup to 648 hours postdose
  Metabolite profiling in plasma, urine, and feces will be performed by liquid chromatography with radiodetection (radio-high performance liquid chromatography [HPLC]) methods. A scintillation counter and/or AMS will be used to detect radioactivity. If needed, plasma and feces samples will be treated with cysteine and/or other reagents before radio-HPLC analyses.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Covance Clinical Research Unit Inc., Madison, Wisconsin
  - Covance Laboratories, Madison, Wisconsin